CLINICAL TRIAL: NCT00080197
Title: An Open-Label Phase II Study of E7070 in Metastatic Breast Cancer Patients Previously Treated With an Anthracycline, a Taxane, and Capecitabine
Brief Title: Study to Evaluate the Efficacy, Safety, and Tolerability of E7070 in Metastatic Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7070-A001-211
Record Dates: First submitted 2004-03-24; First posted 2004-03-25 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2006-10

CONDITIONS: Breast Neoplasms; Metastases
Keywords: Breast Cancer; Cancer of the Breast
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — N-(3-chloro-7-indolyl)-1,4-benzenedisulphonamide

INTERVENTIONS:
Drug: E7070

SUMMARY:
The purpose of this study is to determine if E7070 is an efficacious, safe, and tolerable treatment for patients with metastatic breast cancer who have failed, or could not tolerate, prior treatments with an anthracycline, a taxane, and capecitabine.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be female,
* Patients must have histologically or cytologically confirmed metastatic breast cancer,
* Patients must either have tumors that are resistant/refractory to chemotherapy with an anthracycline, a taxane, capecitabine, and appropriate Herceptin therapy, or tumors that cannot be treated with these agents due to patient's treatment toxicity; therefore, patients must have received 2 prior chemotherapies but no more than 3 prior chemotherapies in the metastatic setting,
* Patients must have at least one uni-dimensionally measurable lesion according to the RECIST criteria in at least one site that has not been irradiated,
* Patients must be aged >= 18 years,
* Patients must have a Karnofsky Performance Status of >= 70%,
* Patients must have a life expectancy of >= 3 months,
* Patients must have adequate renal function as evidenced by serum creatinine <= 1.5 mg/dL, or if > 1.5 but <= 1.8 mg/dL, then a creatinine clearance of >= 45 mL/min,
* Patients must have adequate bone marrow function as evidenced by absolute neutrophil count of >= 1.5 x 109/L, hemoglobin >= 9.0 g/dL, and platelet count >= 100 x 109/L,
* Patients must have adequate liver function as evidenced by bilirubin of <= 1.5 times the upper limits of normal (ULN); alkaline phosphatase <= 3 times ULN and alanine transaminase (ALT) and aspartate transaminase (AST) <= 3 times ULN, unless related to liver metastasis, in which case <= 5 x ULN,
* Patients must have serum electrolytes including calcium (corrected for albumin), magnesium, and potassium (corrected) within normal limits,
* Patients must be willing and able to complete the FACT-B questionnaire,
* Patients must be willing and able to comply with the study protocol for the duration of the study, and
* Patients must give written informed consent prior to any study specific screening procedures with the understanding that the patient may withdraw consent at any time without prejudice.

Exclusion Criteria:

* Patients must not have metastatic disease that can be completely surgically resected,
* Patients who received adjuvant taxane must not have experienced disease progression within 12 months of beginning that therapy,
* Patients must not have received chemotherapy, hormonal therapy, or Herceptin within 2 weeks of E7070 treatment start and must have recovered from any chemotherapy-related or other therapy-related toxicity at study entry,
* Patients must not have received investigational drugs including immunotherapy, gene therapy, or other biologic therapy; antineoplastic therapy; or radiation therapy (other than required for palliation of bone pain or chest ulceration) within 2 weeks of E7070 treatment,
* Patients must not have received prior treatment with Mitomycin C or nitrosoureas,
* Patients must not have undergone high dose chemotherapy with hematopoietic stem cell rescue,
* Patients must not have untreated brain metastases (Patients who have been treated for central nervous system (CNS) metastases must be asymptomatic and radiologically stable [not receiving radiation] and must not have been receiving steroids for 4 weeks prior to entry.

Patients without known CNS metastases who are symptomatic for CNS metastasis must be evaluated with a CT scan or MRI scan prior to E7070 treatment.),

* Patients must not have had major surgery without full recovery within 4 weeks of E7070 treatment start,
* Patients must not have pulmonary lymphatic involvement that results in pulmonary dysfunction requiring active treatment, including the use of oxygen,
* Patients must not have leptomeningeal metastasis,
* Patients must not have evidence of clinically relevant ascites or pleural effusion requiring more than one isolated paracentesis or pleurocentesis per month prior to study start,
* Patients must not be expected to require more than one isolated paracentesis or pleurocentesis per month during the study for the treatment of clinically relevant ascites or pleural effusion,
* Patients must not be pregnant or breast-feeding and must practice adequate contraception if not surgically sterile,
* Patients must not have severe medically uncontrolled intercurrent illness/infection,
* Patients must not have had unstable angina or myocardial infarction in the past 6 months,
* Patients must not have serious cardiac arrhythmia or symptomatic congestive heart failure >= Grade II (NYHA classification),
* Patients must not have a history of prolonged QT, QTc > 470 ms (Bazett's correction) at entry, or history of torsade de pointes,
* Patients must not have recent history (<= 12 months) of active or chronic viral hepatitis,
* Patients must not have organ allografts,
* Patients must not have known history of HIV positivity,
* Patients must not have a history of hypersensitivity to sulfonamides,
* Patients must not have a history of uncontrolled seizures,
* Patients must not have had a prior malignancy, other than carcinoma in situ of the cervix or nonmelanoma skin cancer, unless the prior malignancy was diagnosed and definitively treated >= 5 years previously with no subsequent evidence of recurrence, or
* Patients must not have other significant disease or disorders that, in the Investigator's opinion, would exclude the patient from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2004-02; Study Completion 2005-05

PRIMARY OUTCOMES:
Objective Response Rate

SECONDARY OUTCOMES:
Duration of Response
Time-to-Progression
Overall Survival
Safety
Tolerability
Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Silberman, M.D., Study Director — Eisai Inc.
Locations (35):
- United States (34):
  - Birmingham, Alabama
  - Hoover, Alabama
  - Sedona, Arizona
  - Denver, Colorado
  - Torrington, Connecticut
  - Fort Myers, Florida
  - Ocoee, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Skokie, Illinois
  - Urbana, Illinois
  - Indianapolis, Indiana
  - Overland Park, Kansas
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Albany, New York
  - Winston-Salem, North Carolina
  - Kettering, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Clairton, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Wexford, Pennsylvania
  - Greenville, South Carolina
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Fredericksburg, Texas
  - Houston, Texas
  - Irving, Texas
  - Tyler, Texas
  - Fairfax, Virginia
  - Spokane, Washington
  - Vancouver, Washington
- Edmonton, Alberta, Canada

REFERENCES:
- See also: Related Info — http://www.eisai.com